CLINICAL TRIAL: NCT00463164
Title: Functional MRI of Cognitive Control in Autism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Other Study IDs: 06-179
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Autism
Keywords: functional MRI
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the role of fronto-striatal circuits and cognitive control in the perseverative and inflexible behavior that is a defining feature of autism. We hypothesize that deficits in the development of fronto-striatal circuitry may underlie cognitive inflexibility in autism. Specifically, we hypothesize that repetitive, inflexible behavior arises as (1) fronto-striatal systems are capable of learning patterns present in the environment (as in implicit learning paradigms), but are unable to adapt behavior to changing circumstances, related to either (2) decreased ability of basal ganglia to detect violations of expectancy, (3) decreased ability of prefrontal cortex to respond to detected violations, or (4) decreased connectivity of the circuits. We are conducting three functional Magnetic Resonance Imaging (fMRI) studies to address these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 - 12 years at inclusion

Inclusion criteria for subjects with autism

* DSM-IV (APA, 1994) diagnosis of autism, according to ADI-R interview

Inclusion criteria for controls

* No DSM-IV (APA, 1994) diagnosis, according to DISC interview
* No scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)
* IQ > 70

Exclusion Criteria:

* Major illness of the cardiovascular, the endocrine, the pulmonal or the gastrointestinal system
* Presence of metal objects in or around the body (pacemaker, dental braces)
* History of or present neurological disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90
Dates: Start 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Durston, Ph.D., Principal Investigator — Rudolf Magnus Institute of Neuroscience, University Medical Center Utrecht; Herman van Engeland, M.D. Ph.D., Study Chair — Rudolf Magnust Institute of Neuroscience, UMC Utrecht
Locations (1):
- Dept. of Child and Adolescent Psychiatry, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Lab homepage with info for subjects (in Dutch) — http://www.niche-lab.nl